CLINICAL TRIAL: NCT00340873
Title: Molecular Epidemiology of Dioxin-Related Illness in Seveso
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999995038; OH95-C-N038
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: 2,3,7,8-Tetrachlorodibenzo-Para-Dioxin (TCDD) Exposure
Keywords: Molecular Epidemiology; Cross-Sectional; Gene-Enviroment Interaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Cases: Individuals exposed to digoxin
- Controls: Individuals not exposed to digoxin

SUMMARY:
In 1976 an accidental explosion in a chemical plant 16 miles north of Milan resulted in contamination of the local population with 2, 3, 7, 8-terachlorodibenzo-para-dioxin (TCDD). There is evidence that TCDD and related phenoxy herbicides act as teratogens, tumor promoters, and carcinogens in experimental animals. In human, TCDD causes chloracne in those exposed. Associations with various cancers have been reported, but the precise role in human toxicity, immune and reproductive dysfunction, and cancer is controversial.

The Seveso accident provides a unique opportunity for an epidemiological investigation in that the exposures are the highest recorded in humans, the exposure involves TCDD without other contaminants, and a cohort in the involved and surrounding area has been enumerated.

There is inter-individual variation in the action of genes involved in TCDD effect in human cells. The quality of human AH receptor, and the CYP1A1 and arnt genotypes are examples of susceptibility markers that may identify subjects at high risk for TCDD-related disease. A hypothesis that could explain the inconsistent association of TCDD exposure with cancer is that genetic susceptibility may influence which individuals are adversely affected by TCDD exposure.

The study is proceeding in three phases. The first is a pilot/validation study that is complete (field activities) and involved 126 subjects. The second is a case-control study of about 100 individuals with chloracne and 100 controls. The field components of phase one and two are complete, and analyses of results are underway. The third and final phase is a planned case-control study of TCDD-related cancers that will include approximately 125 cases and 125 controls.

The study includes a questionnaire/interview and a biospecimen collection; 73 ml of blood are obtained from each participant.

DETAILED DESCRIPTION:
In 1976 an accidental explosion in a chemical plant 16 miles north of Milan resulted in contamination of the local population with 2, 3, 7, 8-tetrachlorodibenzo-para-dioxin (TCDD). There is evidence that TCDD and related phenoxy herbicides act as teratogens, tumor promoters, and carcinogens in experimental animals. In human, TCDD causes chloracne in those exposed. Associations with various cancers have been reported, but the precise role in human toxicity, immune and reproductive dysfunction, and cancer is controversial.

The Seveso accident provides a unique opportunity for an epidemiological investigation in that the exposures are the highest recorded in humans, the exposure involves TCDD without other contaminants, and a cohort in the involved and surrounding area has been enumerated.

There is inter-individual variation in the action of genes involved in TCDD effect in human cells. The quality of human AH receptor, and the CYP1A1 and arnt genotypes are examples of susceptibility markers that may identify subjects at high risk for TCDD-related disease. A hypothesis that could explain the inconsistent association of TCDD exposure with cancer is that genetic susceptibility may influence which individuals are adversely affected by TCDD exposure.

The study is in three phases. The first is a pilot/validation study of 126 highly exposed and not exposed subjects. The second is a case-control study of 100 individuals with chloracne and 100 controls. The field components of phase one and two are complete. The third and final phase is a planned case-control study of TCDD-related cancers that will include approximately 125 cases and 125 controls.

Using different methods to estimate TCDD levels below the detection limit, we found that, approximately 20 years after the accident, plasma TCDD was still elevated in subjects from the exposed areas, particularly in women, and was negatively associated with IgG plasma levels. Subjects who developed chloracne after the accident had high TCDD levels, and no evidence of TCDD-related long-term toxicity.

The analyses of the expression of key genes in the aryl hydrocarbon receptor (AhR) pathway, which is necessary for most TCDD effects, showed a significant reduction in AhR expression by increasing plasma dioxin levels. Cytochrome P450 gene SNPs and haplotypes were associated with variable TCDD-related gene inducibility.

On-going studies are examining the proteomics and gene expression pattern (by microarray) in exposed subjects compared with not exposed individuals, and the frerquency of t(14;18) translocations in lymphocytes from the same subjects.

The study includes a questionnaire/interview and a biospecimen collection; 73 ml of blood were obtained from each participant.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects exposed to TCDD in the region of Lombardy, Italy.

EXCLUSION CRITERIA:

1. severe medical illness: liver (cirrhosis [based on medical history], chronic or acute hepatitis [based on transaminase elevation, SGOT greater than 200 IU or SGPT greater than 200 IU]), kidney (hemo- or peritoneal dialysis dependent), cardiac (myocardial infarct in the last 6 months), AIDS (or known HIV positive), major psychiatric illness (decompensated schizophrenia);
2. IV drug abuse;
3. individuals receiving a few specific medications known to interfere with specific assays (i.e., phenobarbitol), other medication use will be recorded;
4. non-Italian origin;
5. Any condition which precludes obtaining informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included subjects who were exposed to dioxin and controls not exposed to dioxin.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 1994-12-12 (Actual); Primary Completion 2007-08-13 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
To determine the effect of TCDD exposure on human health | Ongoing
  Cancer Risk

CONTACTS AND LOCATIONS:
Overall Officials: Maria T Landi, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- University of Milan, Milan, Italy

REFERENCES:
- [Background] Baccarelli A, Giacomini SM, Corbetta C, Landi MT, Bonzini M, Consonni D, Grillo P, Patterson DG, Pesatori AC, Bertazzi PA. Neonatal thyroid function in Seveso 25 years after maternal exposure to dioxin. PLoS Med. 2008 Jul 29;5(7):e161. doi: 10.1371/journal.pmed.0050161. PMID 18666825
- [Background] Consonni D, Sindaco R, Agnello L, Caporaso NE, Landi MT, Pesatori AC, Bertazzi PA. Plasma levels of dioxins, furans, non-ortho-PCBs, and TEQs in the Seveso population 17 years after the accident. Med Lav. 2012 Jul-Aug;103(4):259-67. PMID 22880488
- [Background] McHale CM, Zhang L, Hubbard AE, Zhao X, Baccarelli A, Pesatori AC, Smith MT, Landi MT. Microarray analysis of gene expression in peripheral blood mononuclear cells from dioxin-exposed human subjects. Toxicology. 2007 Jan 5;229(1-2):101-13. doi: 10.1016/j.tox.2006.10.004. Epub 2006 Oct 17. PMID 17101203